CLINICAL TRIAL: NCT01147016
Title: A Phase II Study of Anti-CD3 x Anti-HER2/Neu (Her2Bi) Armed Activated T Cells (ATC) After Neoadjuvant Chemotherapy in Women With HER2/Neu (0-2+), Hormone Receptor (HR) Negative Stage II-III Breast Cancers
Brief Title: Targeted T Cells After Neoadjuvant Chemotherapy in Treating Women With Stage II or III Breast Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary co-investigator leaving the institution & funding transfer.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abhinav Deol, Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-056(b); P30CA022453 (NIH); WSU-2010-056 (Other: Barbara Ann Karmanos Institute); NCT01658969 (obsolete NCT alias)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-negative breast cancer; HER2-negative breast cancer; male breast cancer; progesterone receptor-negative breast cancer; recurrent breast cancer; stage IIA breast cancer; stage IIB breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; Albumin-Bound Paclitaxel; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HER2Bi-armed activated T cells + Neoadjuvant Chemotherapy (Experimental): HER2Bi-armed activated T cells - Total of 4 of the T cell infusions IV over a period of 1 month
  Cyclophosphamide, doxorubicin hydrochloride, paclitaxel -As prescribed by physician, standard of care.
  Interventions: Biological: HER2Bi-armed activated T cells; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Other: laboratory biomarker analysis; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Biological: HER2Bi-armed activated T cells — Total of 4 of the T cell infusions intravenously over a period of 1 month.
Drug: cyclophosphamide — As prescribed by physician, standard of care.
  Other Names: Cytoxan®
Drug: doxorubicin hydrochloride — As prescribed by physician, standard of care.
  Other Names: Adriamycin®; Rubex®
Drug: paclitaxel — As prescribed by physician, standard of care.
  Other Names: Abraxane®; Onxol®; Taxol
Other: laboratory biomarker analysis — Immune studies will be done pre-immunotherapy, prior to the third infusion of activated T-cells, at the time of surgery, and 1 month after immunotherapy. If there are positive findings, additional optional studies will be done at 3, 6, and 12 months, if the immune studies show changes worthy of follow-up studies.
Procedure: neoadjuvant therapy — As prescribed by physician, standard of care.
Procedure: therapeutic conventional surgery — As recommended by physician, post immunotherapy.

SUMMARY:
RATIONALE: Neoadjuvant chemotherapy for women with stage II-III Her negative breast cancer followed by Her2Bi armed activated T cells (ATCs) may significantly improve the pathologic complete response (pCR) rate at the time of surgery. Arming ex vivo expanded T cells in the laboratory may help the T cells kill more tumor cells when they are put back in the body. Giving combination neoadjuvant chemotherapy followed by laboratory-treated T cells before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II clinical trial is studying how well giving laboratory-treated T cells after neoadjuvant chemotherapy works in treating women with stage II or stage III breast cancer undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate progression-free survival (PFS) in women with stage II-III triple-negative breast cancer without a complete pathologic response (cPR) who receive a regimen of neoadjuvant chemotherapy (chemoT), surgery, and/or irradiation followed by 8 infusions of ~10-15 x 10^9 Her2Bi-armed activated T cells (ATC) (aATC) given twice per week for 4 weeks in combination with IL-2 (aldesleukin) (300,000 IU/m^2/day) and GM-CSF (sargramostim) (250 μg/m^2/twice per week) beginning 3 days before the 1st infusion and ending 1 week after the last infusion (defined as immunotherapy).

II. To estimate the change from baseline (pre immunotherapy [IT]) to post-IT in specific cytotoxicity and interferon gamma (IFN-γ) enzyme-linked immunosorbent spots (Elispots) of lymphocytes in the blood directed at breast cancer cells.

III. To investigate if pathologic response and the changes in numbers and proportion of infiltrating cells and cancer stem cells in the tumor at the time of surgery are associated with progressive disease.

OUTLINE:

NEOADJUVANT CHEMOTHERAPY: Patients receive dose-dense AC-T regimen comprising doxorubicin hydrochloride intravenously (IV) and cyclophosphamide IV once every 2 weeks for 4 courses followed by paclitaxel IV once every 2 weeks for 4 courses or paclitaxel IV once weekly for 12 weeks. Or, patients receive TAC regimen comprising docetaxel IV, doxorubicin hydrochloride IV, and cyclophosphamide IV once every 3 weeks for 6 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.

IMMUNOTHERAPY: Beginning 3 weeks after the last dose of chemotherapy, patients receive Her2Bi-armed activated T cells IV over 5-30 minutes twice weekly for 4 weeks. Patients also receive aldesleukin subcutaneously (SC) daily beginning 3 days before the first T cell infusion and ending 1 week after the last infusion.

SURGERY: Patients then undergo surgical resection of the breast 2 weeks later.

After completion of study treatment, patients may be followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria

* Signed and dated institutional review board (IRB)-approved consent form
* Women of reproductive potential must agree to use an effective nonhormonal method of contraception during therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 and/or Karnofsky PS of >= 70%
* Diagnosis of invasive adenocarcinoma of the breast made by core needle biopsy
* Palpable primary breast tumor measuring >= 2.0 cm on physical exam or imaging prior to neoadjuvant chemotherapy
* Patients with stage II-IIIB breast cancer that is HER2-negative by immunohistochemistry (IHC) (0-2+) and fluorescence in situ hybridization (FISH) (HER2/chromosome enumeration probe [CEP]17 amplification ratio < 2.0) who have completed "third generation" neoadjuvant chemoT and planned local treatment (surgery and radiation if indicated); estrogen receptor (ER) or progesterone receptor (PR) status should be negative
* Patients may have lymph node positive or negative disease, as long as they have clinical/pathologic stage II or IIIB breast cancer; patients may have the lymph nodes assessed by any method deemed appropriate by the treating physicians, including pre-neoadjuvant therapy sentinel lymph node biopsy
* Presence of residual disease measuring at least 5mm (as single foci or in aggregate) on final pathology following surgery
* Patients must discontinue sex hormone therapy prior to registration, e.g. birth control pills, hormonal replacement therapy
* Absolute neutrophil count (ANC) must be >= 1000/mm^3
* Platelet count must be >= 100,000/mm^3
* Hemoglobin must be >= 9.0 mg/dL
* Total bilirubin must be =< the upper limit of normal (ULN) for the lab unless the patient has a grade 1 bilirubin elevation (> ULN to 1.5 x ULN) resulting from Gilbert's disease or similar syndrome due to slow conjugation of bilirubin; and
* Alkaline phosphatase must be =< 2.5 x ULN for the lab
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) must be =< 1.5 x ULN for the lab
* Alkaline phosphatase and AST/ALT may not both be > the ULN; for example, if the alkaline phosphatase is > the ULN but =< 2.5 x ULN, then the AST/ALT must be =< the ULN; if the AST/ALT is > the ULN but =< 1.5 x ULN, then the alkaline phosphatase must be =< ULN
* Patients with either skeletal pain or alkaline phosphatase that is > ULN must have a bone scan showing they do not have metastatic disease; suspicious findings on bone scan must be confirmed as benign by x-ray, magnetic resonance imaging (MRI), or biopsy
* Patients with AST/ALT or alkaline phosphatase > ULN must have liver imaging that does not demonstrate metastatic disease
* Patients with AST/ALT > ULN must have negative hepatitis studies
* Patients with stage II disease and clinical suspicion for metastatic disease based on reported symptoms, physical examination findings, or laboratory abnormalities must have staging studies demonstrating no evidence of metastatic disease (with exception of axillary lymph nodes or mammary nodes); patients with stage IIIA disease must have staging studies demonstrating no evidence of metastatic disease (with exception of axillary lymph nodes or mammary nodes), even if asymptomatic with normal physical examination and laboratory values; such staging studies must include: chest imaging (chest X-ray, computed tomography [CT], or MRI), abdominal/pelvis imaging (CT or MRI), and bone imaging (bone scan or positron emission tomography [PET]-scan); abnormalities that are indeterminate and too small to biopsy should be followed with further imaging, as appropriate, but do not exclude patients from the study; abnormalities that are suspicious and large enough to biopsy exclude patients from the study, unless a biopsy is performed and is negative for metastatic disease
* Serum creatinine =< 1.5 x ULN for the lab
* Pre-entry core biopsy with sufficient material for correlative studies
* Left Ventricular Ejection Fraction (LVEF) >= 45 % (by multigated acquisition scan [MUGA] or echocardiography)

Exclusion Criteria

* Tumor determined to be HER2-positive by immunohistochemistry (3+) or by fluorescent in situ hybridization (HER2/CEP17 amplification ratio >= 2.0)
* Tumors clinically staged as anyT with N3 disease or unresectable disease
* Evidence of disease progression on neoadjuvant chemo T
* Definitive evidence of metastatic disease with exception of axillary lymph nodes or mammary nodes
* Synchronous bilateral breast cancer (invasive or ductal carcinoma in situ [DCIS])
* Treatment with biotherapy, and/or hormonal therapy for the currently diagnosed breast cancer prior to study entry
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. within 2 weeks prior to the collection of cells
* Prior history of invasive breast cancer (patients with a history of DCIS or lobular carcinoma in situ [LCIS] are eligible)
* Other malignancies unless the patient is considered to be disease-free for 5 or more years prior to randomization and is deemed by the physician to be at low risk for recurrence; patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell or squamous cell carcinoma of the skin
* Known cardiac disease which precludes their ability to receive planned treatments:

  * Angina pectoris that requires the use of anti-anginal medication
  * History of documented congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Severe conduction abnormality
  * Valvular disease with documented cardiac function compromise; and
  * Uncontrolled hypertension defined as blood pressure (BP) that is consistently > 150/90 on antihypertensive therapy at the time of registration (Patients with hypertension that is well controlled on medication are eligible)
* History of myocardial infarction (MI) documented by elevated cardiac enzymes with persistent regional wall motion abnormality on assessment of left ventricular (LV) function (patients with history of MI must have an echo instead of/in addition to a MUGA to evaluate LV wall motion)
* Symptomatic peripheral vascular disease
* Other non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude treatment with any of the treatment regimens or would prevent required follow-up
* Chronic ongoing oral steroid use at the time of registration for any condition (such as asthma, rheumatoid arthritis, etc)
* Administration of any investigational agents within 30 days before study entry
* Pregnancy or lactation at the time of registration
* Psychiatric or addictive disorders or other conditions that in the opinion of the investigators would preclude the patient from complying with the study protocol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-07; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Weise, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated: Single group study
Period: Overall Study
Arm/Group | Treated
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treated
Number analyzed (Participants) | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.5 [39 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
enrollment [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesion
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 years..
Population: Women with stage II-III, HER2/neu (0-2+) negative breast cancer treated with anti-CD3 x anti-HER2neu (Her2BI) armed, activated T cells after neoadjuvant chemotherapy
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Activated T Cells: All participants enrolled
Arm/Group | Activated T Cells
Number analyzed (Participants) | 8
months | 43 [2 to NA] — The sample size is very small and there are too few events to estimate the upper 95% CI.

2. Secondary Outcome: Overall Deaths
Description: Total number of deaths
Time Frame: From date of randomization until date of death from any cause or end of study, whichever came first, assessed up to 7 years
Population: The participant who died had the longest follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 7 years.
Groups:
- Treated: All 8 participants enrolled
Arm/Group | Treated
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treated (N=8)
Hypertension (Cardiac disorders) | 1/1 (1) — Grade 2
chills/rigors (General disorders) | 7 (7) — grade 1 1 grade 2 5 grade 31
Nausea (Gastrointestinal disorders) | 7 (7) — Grade 1 5 Grade 2 1
Vomiting (Gastrointestinal disorders) | 4 (4) — Grade 1 3 Grade 2 1
fatigue (General disorders) | 7 (7) — Grade 1 4 Grade 2 3
Rash (General disorders) | 3 (3) — Grade 1 3
edema (General disorders) | 2 (2) — Grade 1 1 Grade 2 1
neuroppathy (Nervous system disorders) | 3 (3) — Grade 1 1 Grade 2 1 Grade 3 1
hypotension (General disorders) | 5 (5) — Grade 2 5
fever (General disorders) | 6 (6) — grade 1 4 Grade 2 2
hyponatremia (General disorders) | 1 (1) — Grade 1 1
hypoglycemia (Endocrine disorders) | 2 (2) — Grade 1 2
neutropenia (General disorders) | 4 (4) — Grade 1 1 Grade 2 1 Grade 3 1 Grade 4 1
AST elevation (General disorders) | 1 (1) — grade 1 1
ALT elevation (General disorders) | 1 (1) — Grade 1 1
Anemia (Blood and lymphatic system disorders) | 5 (5) — Grade 1 4 Grade 2 1
Afibrillation (Cardiac disorders) | 1 (1) — Grade 2 1
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1 1
Infection (Infections and infestations) | 3 (3) — Grade 1 2 Grade 2 1
Low platelets (Blood and lymphatic system disorders) | 5 (5) — Grade 1 3 Grade 2 2
hypoalbuminemia (Blood and lymphatic system disorders) | 2 (2) — Grade 1 1 Grade 2 1
Alkaline Phosphatase (Blood and lymphatic system disorders) | 2 (2) — Grade 1 1 Grade 2 1
Hypercalcemia (Blood and lymphatic system disorders) | 2 (2) — Grade 1 2 Grade 2 1
Hypocalcemia (Blood and lymphatic system disorders) | 1/1 (1) — Grade 3 1
hypokalemia (Blood and lymphatic system disorders) | 1 (1) — Grade 1 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT01147016/Prot_SAP_000.pdf